CLINICAL TRIAL: NCT02712905
Title: A Phase 1/2, Open-Label, Dose-Escalation/Dose-Expansion, Safety and Tolerability Study of INCB059872 in Subjects With Advanced Malignancies
Brief Title: An Open-Label, Dose-Escalation/Dose-Expansion Safety Study of INCB059872 in Subjects With Advanced Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategic Business Decision
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 59872-101; 2017-001710-28 (EudraCT Number)
Record Dates: First submitted 2016-02-18; First posted 2016-03-18 (Estimated); Results first posted 2023-06-12 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumors and Hematologic Malignancy
Keywords: Acute myeloid leukemia (AML); myelodysplastic syndrome (MDS); small cell lung cancer (SCLC); myelofibrosis (MF); solid tumor, lysine-specific demethylase 1 (LSD1) inhibitor
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Small Cell Lung Carcinoma; Primary Myelofibrosis | interventions — INCB059872; Tretinoin; Azacitidine; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- INCB059872 (Experimental)
  Interventions: Drug: INCB059872
- INCB059872 in combination with other therapies (Experimental): Initial cohort dose of INCB059872 to evaluate different doses of INCB0599872 in combination with other therapies in the following treatment groups:
  * Combination with all-trans retinoic acid (ATRA) in subjects with relapsed/refractory AML.
  * Combination with azacitidine in subjects with newly diagnosed, treatment-naive AML
  * Combination with nivolumab in subjects with advanced SCLC previously progressed on platinum-based treatment.
  Upon identification of the recommended dose(s) for each treatment combination, expansion cohorts of approximately 30 subjects in each treatment group may begin enrollment to further determine safety, tolerability, efficacy, PK, and PD of the selected dose(s).
  Interventions: Drug: INCB059872; Drug: all-trans retinoic acid (ATRA); Drug: azacitidine; Drug: nivolumab

INTERVENTIONS:
Drug: INCB059872 — Initial cohort dose of INCB059872 monotherapy at the protocol-specified starting dose, with subsequent cohort escalations based on protocol-specific criteria. The recommended dose(s) will be taken forward into expansion cohorts.
  INCB059872 tablets to be administered by mouth.
Drug: all-trans retinoic acid (ATRA)
  Arms: INCB059872 in combination with other therapies
Drug: azacitidine
  Arms: INCB059872 in combination with other therapies
Drug: nivolumab
  Arms: INCB059872 in combination with other therapies

SUMMARY:
This is an open-label, dose-escalation/dose-expansion study of INCB059872 in subjects with advanced malignancies. The study will be conducted in 4 parts. Part 1 (mono therapy dose escalation) will determine the recommended dose(s) of INCB059872 for dose expansion, based on maximum tolerated dose and/or a tolerated pharmacologically active dose. Part 2 (dose expansion) will further determine the safety, tolerability, efficacy, PK, and PD of the selected monotherapy dose(s) in AML/MDS, SCLC, myelofibrosis, Ewing sarcoma, and poorly differentiated neuroendocrine tumors. Part 3 will determine the recommended dose(s) of INCB059872 in combination with azacitadine and all-trans retinoic acid in AML and in combination with nivolumab in SCLC. Part 4 will further determine the safety, tolerability, efficacy, PK, and PD of the selected combination dose(s) in Part 3.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age 18 years or older.
* Presence of measurable disease that has been confirmed by histology or cytology.
* Must not be a candidate for potentially curative therapy or standard-of-care approved therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.

Exclusion Criteria:

* Receipt of anticancer medications, anticancer therapies, or investigational drugs within the defined interval before the first administration of study drug.
* Any unresolved toxicity ≥ Grade 2 from previous anticancer therapy except for stable chronic toxicities (≤ Grade 2) not expected to resolve.
* Laboratory and medical history parameters outside Protocol-defined range.
* Known additional malignancy that is progressing or requires active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Zheng, MD, Study Director — Incyte Corporation
Locations (15):
- United States (11):
  - University of Alabama, Birmingham, Alabama
  - Moores UCSD Cancer Center, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - University of Kansas Center for Research, Inc., Kansas City, Kansas
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University, New York, New York
  - Oregon Health Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Institut Jules Bordet, Brussels, Belgium
- Netherlands (3):
  - Netherland Cancer Institute, Amsterdam
  - VU Medical Center, Amsterdam
  - Erasmus MC, Rotterdam

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled at 12 study sites: 10 in the United States and 1 each in Belgium and the Netherlands.
Groups:
- Group A: INCB059872 Monotherapy; 2 mg QOD: Participants with acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) received oral INB059872 2 milligrams (mg) as monotherapy once every other day (QOD) on a 28-day continuous therapy cycle.
- Group A: INCB059872 Monotherapy; 2 mg QD: Participants with AML or MDS received oral INB059872 2 mg as monotherapy once daily (QD) on a 28-day continuous therapy cycle.
- Group A: INCB059872 Monotherapy; 3 mg QOD: Participants with AML or MDS received oral INB059872 3 mg as monotherapy QOD on a 28-day continuous therapy cycle.
- Group A: INCB059872 Monotherapy; 3 mg QD: Participants with AML or MDS received oral INB059872 3 mg as monotherapy QD on a 28-day continuous therapy cycle.
- Group A: INCB059872 Monotherapy; 4 mg QD: Participants with AML or MDS received oral INB059872 4 mg as monotherapy QD on a 28-day continuous therapy cycle.
- Group A: INCB059872 Monotherapy; 5 mg QD: Participants with AML or MDS received oral INB059872 5 mg as monotherapy QD on a 28-day continuous therapy cycle.
- Group B: INCB059872 Monotherapy; 1 mg QD: Participants with small cell lung cancer (SCLC) and other solid malignancies (e.g., endocrine tumors) received oral INB059872 1 mg as monotherapy QD on a 28-day continuous therapy cycle.
- Group B: INCB059872 Monotherapy; 2 mg QOD: Participants with SCLC and other solid malignancies (e.g., endocrine tumors) received oral INB059872 2 mg as monotherapy QOD on a 28-day continuous therapy cycle.
- Group B: INCB059872 Monotherapy; 2 mg QD: Participants with SCLC and other solid malignancies (e.g., endocrine tumors) received oral INB059872 2 mg as monotherapy QD on a 28-day continuous therapy cycle.
- Group B: INCB059872 Monotherapy; 3 mg QOD: Participants with SCLC and other solid malignancies (e.g., endocrine tumors) received oral INB059872 3 mg as monotherapy QOD on a 28-day continuous therapy cycle.
- Group B: INCB059872 Monotherapy; 3 mg QD: Participants with SCLC and other solid malignancies (e.g., endocrine tumors) received oral INB059872 3 mg as monotherapy QD on a 28-day continuous therapy cycle.
- Group B: INCB059872 Monotherapy; 4 mg QOD: Participants with SCLC and other solid malignancies (e.g., endocrine tumors) received oral INB059872 4 mg as monotherapy QOD on a 28-day continuous therapy cycle.
- Group C: Combination Therapy; INCB059872 2 mg QD + ATRA: Participants with relapsed/refractory AML received oral INCB059872 2 mg QD in combination with all-trans retinoic acid (ATRA) (at a starting dose of 45 mg/meters squared [m^2] per day at 2 evenly divided doses) on a 28-day continuous therapy cycle.
- Group C: Combination Therapy; INCB059872 3 mg QD + ATRA: Participants with relapsed/refractory AML received oral INCB059872 3 mg QD in combination with ATRA (at a starting dose of 45 mg/m^2 per day at 2 evenly divided doses) on a 28-day continuous therapy cycle.
- Group C: Combination Therapy; INCB059872 4 mg QD + ATRA: Participants with relapsed/refractory AML received oral INCB059872 4 mg QD in combination with ATRA (at a starting dose of 45 mg/m^2 per day at 2 evenly divided doses) on a 28-day continuous therapy cycle.
- Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine: Participants with newly diagnosed, treatment-naïve AML or MDS received INCB059872 2 mg QD on a 28-day continuous therapy cycle in combination with azacitidine, administered at a starting dose of 75 mg/m^2 subcutaneously or intravenously for 7 days during the first 9-day period of each 28-day treatment cycle.
- Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine: Participants with newly diagnosed, treatment-naïve AML or MDS received INCB059872 3 mg QD on a 28-day continuous therapy cycle in combination with azacitidine, administered at a starting dose of 75 mg/m^2 subcutaneously or intravenously for 7 days during the first 9-day period of each 28-day treatment cycle.
- Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab: Participants with SCLC received oral INCB059872 3 mg QOD on a 28-day continuous therapy cycle in combination with nivolumab, administered at 3 mg/kilogram (kg) intravenously over 60 minutes every 2 weeks of each 28-day treatment cycle.
Period: Monotherapy
Arm/Group | Group A: INCB059872 Monotherapy; 2 mg QOD | Group A: INCB059872 Monotherapy; 2 mg QD | Group A: INCB059872 Monotherapy; 3 mg QOD | Group A: INCB059872 Monotherapy; 3 mg QD | Group A: INCB059872 Monotherapy; 4 mg QD | Group A: INCB059872 Monotherapy; 5 mg QD | Group B: INCB059872 Monotherapy; 1 mg QD | Group B: INCB059872 Monotherapy; 2 mg QOD | Group B: INCB059872 Monotherapy; 2 mg QD | Group B: INCB059872 Monotherapy; 3 mg QOD | Group B: INCB059872 Monotherapy; 3 mg QD | Group B: INCB059872 Monotherapy; 4 mg QOD | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab
Started | 3 | 6 | 1 | 5 | 18 | 2 | 3 | 3 | 1 | 36 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 1 | 5 | 18 | 2 | 3 | 3 | 1 | 36 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 5 | 0 | 3 | 15 | 1 | 3 | 3 | 0 | 27 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 4 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Started New Cancer Drug | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Combination Therapy
Arm/Group | Group A: INCB059872 Monotherapy; 2 mg QOD | Group A: INCB059872 Monotherapy; 2 mg QD | Group A: INCB059872 Monotherapy; 3 mg QOD | Group A: INCB059872 Monotherapy; 3 mg QD | Group A: INCB059872 Monotherapy; 4 mg QD | Group A: INCB059872 Monotherapy; 5 mg QD | Group B: INCB059872 Monotherapy; 1 mg QD | Group B: INCB059872 Monotherapy; 2 mg QOD | Group B: INCB059872 Monotherapy; 2 mg QD | Group B: INCB059872 Monotherapy; 3 mg QOD | Group B: INCB059872 Monotherapy; 3 mg QD | Group B: INCB059872 Monotherapy; 4 mg QOD | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 1 | 7 | 1 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 1 | 7 | 1 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 1 | 3 | 1 | 3
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Unknown; Did Not Complete End of Study Case Report Form Prior to Site Closure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: INCB059872 Monotherapy; 2 mg QOD | Group A: INCB059872 Monotherapy; 2 mg QD | Group A: INCB059872 Monotherapy; 3 mg QOD | Group A: INCB059872 Monotherapy; 3 mg QD | Group A: INCB059872 Monotherapy; 4 mg QD | Group A: INCB059872 Monotherapy; 5 mg QD | Group B: INCB059872 Monotherapy; 1 mg QD | Group B: INCB059872 Monotherapy; 2 mg QOD | Group B: INCB059872 Monotherapy; 2 mg QD | Group B: INCB059872 Monotherapy; 3 mg QOD | Group B: INCB059872 Monotherapy; 3 mg QD | Group B: INCB059872 Monotherapy; 4 mg QOD | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab | Total
Number analyzed (Participants) | 3 | 6 | 1 | 5 | 18 | 2 | 3 | 3 | 1 | 36 | 3 | 7 | 5 | 7 | 1 | 7 | 1 | 6 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (5.20) | 58.0 (9.53) | NA (NA) — Unable to report age for a single participant due to privacy concerns. | 57.4 (21.93) | 63.8 (12.02) | 51.0 (18.38) | 46.3 (22.59) | 63.0 (17.09) | NA (NA) — Unable to report age for a single participant due to privacy concerns. | 57.8 (13.95) | 51.0 (11.53) | 63.0 (4.86) | 61.0 (9.19) | 63.6 (13.83) | NA (NA) — Unable to report age for a single participant due to privacy concerns. | 73.4 (9.02) | NA (NA) — Unable to report age for a single participant due to privacy concerns. | 68.7 (9.48) | 60.8 (13.39)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: For treatment arms in which a single participant was enrolled, data have not been reported due to privacy concerns (denoted Number Analyzed=0 for treatment arm).
  Participants
    number analyzed (Participants) | 3 | 6 | 0 | 5 | 18 | 2 | 3 | 3 | 0 | 36 | 3 | 7 | 5 | 7 | 0 | 7 | 0 | 6 | 111
    Female | 3 | 3 |  | 3 | 9 | 2 | 1 | 3 |  | 16 | 0 | 4 | 0 | 4 |  | 3 |  | 3 | 54
    Male | 0 | 3 |  | 2 | 9 | 0 | 2 | 0 |  | 20 | 3 | 3 | 5 | 3 |  | 4 |  | 3 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: For treatment arms in which a single participant was enrolled, data have not been reported due to privacy concerns (denoted Number Analyzed=0 for treatment arm).
  Participants
    number analyzed (Participants) | 3 | 6 | 0 | 5 | 18 | 2 | 3 | 3 | 0 | 36 | 3 | 7 | 5 | 7 | 0 | 7 | 0 | 6 | 111
    Hispanic or Latino | 0 | 1 |  | 0 | 2 | 1 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 |  | 0 |  | 0 | 4
    Not Hispanic or Latino | 3 | 5 |  | 5 | 16 | 1 | 3 | 3 |  | 36 | 3 | 7 | 5 | 7 |  | 7 |  | 6 | 107
    Unknown or Not Reported | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 |  | 0 |  | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: For treatment arms in which a single participant was enrolled, data have not been reported due to privacy concerns (denoted Number Analyzed=0 for treatment arm).
  Participants
    White: number analyzed (Participants) | 3 | 6 | 0 | 5 | 18 | 2 | 3 | 3 | 0 | 36 | 3 | 7 | 5 | 7 | 0 | 7 | 0 | 6 | 111
    White | 3 | 4 |  | 4 | 15 | 2 | 2 | 2 |  | 31 | 3 | 6 | 5 | 6 |  | 7 |  | 6 | 96
    Black or African American: number analyzed (Participants) | 3 | 6 | 0 | 5 | 18 | 2 | 3 | 3 | 0 | 36 | 3 | 7 | 5 | 7 | 0 | 7 | 0 | 6 | 111
    Black or African American | 0 | 2 |  | 0 | 1 | 0 | 0 | 1 |  | 3 | 0 | 1 | 0 | 0 |  | 0 |  | 0 | 8
    Asian: number analyzed (Participants) | 3 | 6 | 0 | 5 | 18 | 2 | 3 | 3 | 0 | 36 | 3 | 7 | 5 | 7 | 0 | 7 | 0 | 6 | 111
    Asian | 0 | 0 |  | 0 | 0 | 0 | 1 | 0 |  | 1 | 0 | 0 | 0 | 0 |  | 0 |  | 0 | 2
    American-Indian/Alaska Native: number analyzed (Participants) | 3 | 6 | 0 | 5 | 18 | 2 | 3 | 3 | 0 | 36 | 3 | 7 | 5 | 7 | 0 | 7 | 0 | 6 | 111
    American-Indian/Alaska Native | 0 | 0 |  | 0 | 1 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 |  | 0 |  | 0 | 1
    Non-White: number analyzed (Participants) | 3 | 6 | 0 | 5 | 18 | 2 | 3 | 3 | 0 | 36 | 3 | 7 | 5 | 7 | 0 | 7 | 0 | 6 | 111
    Non-White | 0 | 0 |  | 1 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 |  | 0 |  | 0 | 1
    Unknown/Not Specified: number analyzed (Participants) | 3 | 6 | 0 | 5 | 18 | 2 | 3 | 3 | 0 | 36 | 3 | 7 | 5 | 7 | 0 | 7 | 0 | 6 | 111
    Unknown/Not Specified | 0 | 0 |  | 0 | 1 | 0 | 0 | 0 |  | 1 | 0 | 0 | 0 | 0 |  | 0 |  | 0 | 2
    Declined to Report: number analyzed (Participants) | 3 | 6 | 0 | 5 | 18 | 2 | 3 | 3 | 0 | 36 | 3 | 7 | 5 | 7 | 0 | 7 | 0 | 6 | 111
    Declined to Report | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 1 |  | 0 |  | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Receiving INCB059872 Monotherapy With Any Treatment-emergent Adverse Event (TEAE)
Description: Adverse events (AEs) were defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study drug(s). TEAEs were defined as AEs either reported for the first time or the worsening of pre-existing events after the first dose of study drug and within 30 days of the last administration of study drug.
Time Frame: up to 588 days
Population: Safety Population: all enrolled participants who received at least 1 dose of INCB059872, ATRA, azacitidine, or nivolumab
Measure: Count of Participants; unit: Participants
Groups:
- Group A: INCB059872 Monotherapy; 2 mg QOD: Participants with acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) received INB059872 2 milligrams (mg) as monotherapy once every other day (QOD) on a 28-day continuous therapy cycle.
- Group A: INCB059872 Monotherapy; 2 mg QD: Participants with AML or MDS received INB059872 2 mg as monotherapy once daily (QD) on a 28-day continuous therapy cycle.
- Group A: INCB059872 Monotherapy; 3 mg QOD: Participants with AML or MDS received INB059872 3 mg as monotherapy QOD on a 28-day continuous therapy cycle.
- Group A: INCB059872 Monotherapy; 3 mg QD: Participants with AML or MDS received INB059872 3 mg as monotherapy QD on a 28-day continuous therapy cycle.
- Group A: INCB059872 Monotherapy; 4 mg QD: Participants with AML or MDS received INB059872 4 mg as monotherapy QD on a 28-day continuous therapy cycle.
- Group A: INCB059872 Monotherapy; 5 mg QD: Participants with AML or MDS received INB059872 5 mg as monotherapy QD on a 28-day continuous therapy cycle.
- Group B: INCB059872 Monotherapy; 1 mg QD: Participants with small cell lung cancer (SCLC) and other solid malignancies (e.g., endocrine tumors) received INB059872 1 mg as monotherapy QD on a 28-day continuous therapy cycle.
- Group B: INCB059872 Monotherapy; 2 mg QOD: Participants with SCLC and other solid malignancies (e.g., endocrine tumors) received INB059872 2 mg as monotherapy QOD on a 28-day continuous therapy cycle.
- Group B: INCB059872 Monotherapy; 2 mg QD: Participants with SCLC and other solid malignancies (e.g., endocrine tumors) received INB059872 2 mg as monotherapy QD on a 28-day continuous therapy cycle.
- Group B: INCB059872 Monotherapy; 3 mg QOD: Participants with SCLC and other solid malignancies (e.g., endocrine tumors) received INB059872 3 mg as monotherapy QOD on a 28-day continuous therapy cycle.
- Group B: INCB059872 Monotherapy; 3 mg QD: Participants with SCLC and other solid malignancies (e.g., endocrine tumors) received INB059872 3 mg as monotherapy QD on a 28-day continuous therapy cycle.
- Group B: INCB059872 Monotherapy; 4 mg QOD: Participants with SCLC and other solid malignancies (e.g., endocrine tumors) received INB059872 4 mg as monotherapy QOD on a 28-day continuous therapy cycle.
Arm/Group | Group A: INCB059872 Monotherapy; 2 mg QOD | Group A: INCB059872 Monotherapy; 2 mg QD | Group A: INCB059872 Monotherapy; 3 mg QOD | Group A: INCB059872 Monotherapy; 3 mg QD | Group A: INCB059872 Monotherapy; 4 mg QD | Group A: INCB059872 Monotherapy; 5 mg QD | Group B: INCB059872 Monotherapy; 1 mg QD | Group B: INCB059872 Monotherapy; 2 mg QOD | Group B: INCB059872 Monotherapy; 2 mg QD | Group B: INCB059872 Monotherapy; 3 mg QOD | Group B: INCB059872 Monotherapy; 3 mg QD | Group B: INCB059872 Monotherapy; 4 mg QOD
Number analyzed (Participants) | 3 | 6 | 1 | 5 | 18 | 2 | 3 | 3 | 1 | 36 | 3 | 7
Participants | 3 | 6 | 1 | 5 | 18 | 2 | 3 | 3 | 1 | 36 | 3 | 7

2. Primary Outcome: Number of Participants Receiving INCB059872 Combination Therapy With Any TEAE
Description: AEs were defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or required changes in the study drug(s). TEAEs were defined as AEs either reported for the first time or the worsening of pre-existing events after the first dose of study drug and within 30 days of the last administration of study drug.
Time Frame: up to 1387 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Group C: Combination Therapy; INCB059872 2 mg QD + ATRA: Participants with relapsed/refractory AML received INCB059872 2 mg QD in combination with all-trans retinoic acid (ATRA) (at a starting dose of 45 mg/meters squared [m^2] per day at 2 evenly divided doses) on a 28-day continuous therapy cycle.
Arm/Group | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab
Number analyzed (Participants) | 5 | 7 | 1 | 7 | 1 | 6
Participants | 5 | 7 | 1 | 7 | 1 | 6

3. Secondary Outcome: Objective Response Rate (ORR) in Participants With the Indicated Type of Solid Tumors Who Received INCB059872 Monotherapy
Description: ORR was defined as the percentage of participants who achieved a best overall response of complete response (CR) or a partial response (PR), per investigator assessment according to Response Evaluation Criteria in Solid Tumors version 1.1 (RESIST v1.1), recorded before and including the first event of progressive disease (PD). CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 millimeters (mm). PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to 518 days
Population: Full Analysis Set: all enrolled participants who received at least 1 dose of INCB059872, ATRA, azacitidine, or nivolumab. Only participants with the indicated type of solid tumor who received monotherapy were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: INCB059872 Monotherapy; 2 mg QOD | Group A: INCB059872 Monotherapy; 2 mg QD | Group A: INCB059872 Monotherapy; 3 mg QOD | Group A: INCB059872 Monotherapy; 3 mg QD | Group A: INCB059872 Monotherapy; 4 mg QD | Group A: INCB059872 Monotherapy; 5 mg QD | Group B: INCB059872 Monotherapy; 1 mg QD | Group B: INCB059872 Monotherapy; 2 mg QOD | Group B: INCB059872 Monotherapy; 2 mg QD | Group B: INCB059872 Monotherapy; 3 mg QOD | Group B: INCB059872 Monotherapy; 3 mg QD | Group B: INCB059872 Monotherapy; 4 mg QOD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 36 | 3 | 7
percentage of participants
  SCLC: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 1 | 3
  SCLC |  |  |  |  |  |  |  |  |  | 0.0 | 0.0 | 0.0
  Ewing's sarcoma: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
  Ewing's sarcoma |  |  |  |  |  |  |  |  |  | 0.0 |  |
  Poorly differentiated neuroendocrine tumors: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 12 | 0 | 0
  Poorly differentiated neuroendocrine tumors |  |  |  |  |  |  | 0.0 |  |  | 0.0 |  |
  Other solid tumors: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 3 | 2 | 4
  Other solid tumors |  |  |  |  |  |  | 0.0 | 0.0 | 0.0 | 0.0 | 50.0 | 0.0

4. Secondary Outcome: ORR for Altering the Natural History of the Disease in Participants With Acute Myeloid Leukemia (AML) Who Received INCB059872 Monotherapy
Description: ORR was defined as the percentage of participants who achieved a best overall response of complete remission or complete remission with incomplete hematologic recovery (CRi), per the International Working Group Response Criteria for AML, recorded before and including the first event of progression (treatment failure, relapse, and PD) based on altering the natural history of the disease. Complete remission: absolute neutrophil count (ANC) ≥1.0 x 10^9/Liter (L), platelet count ≥100 x 10^9/L, bone marrow with less than 5% blast cells, Auer rods not detectable; no platelet, or whole blood transfusions for 7 days prior to the date of the hematology assessment. CRi: complete remission, but the ANC count may be < 1.0 x 10^9/L and/or the platelet count may be <100 x 10^9/L.
Time Frame: up to 85 days
Population: Full Analysis Set. Only participants with AML who received monotherapy were analyzed. The participant in Group A receiving 3 mg QOD was on treatment for less than a week and therefore was not evaluated for efficacy.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: INCB059872 Monotherapy; 2 mg QOD | Group A: INCB059872 Monotherapy; 2 mg QD | Group A: INCB059872 Monotherapy; 3 mg QOD | Group A: INCB059872 Monotherapy; 3 mg QD | Group A: INCB059872 Monotherapy; 4 mg QD | Group A: INCB059872 Monotherapy; 5 mg QD | Group B: INCB059872 Monotherapy; 1 mg QD | Group B: INCB059872 Monotherapy; 2 mg QOD | Group B: INCB059872 Monotherapy; 2 mg QD | Group B: INCB059872 Monotherapy; 3 mg QOD | Group B: INCB059872 Monotherapy; 3 mg QD | Group B: INCB059872 Monotherapy; 4 mg QOD
Number analyzed (Participants) | 3 | 5 | 0 | 4 | 12 | 2 | 0 | 0 | 0 | 0 | 0 | 0
percentage of participants | 0.0 | 0.0 |  | 0.0 | 0.0 | 0.0 |  |  |  |  |  |

5. Secondary Outcome: ORR for Altering the Natural History of the Disease in Participants With Myelodysplastic Syndrome (MDS) Who Received INCB059872 Monotherapy
Description: ORR was defined as the percentage of participants who achieved a best overall response of complete remission, partial remission, or bone marrow complete remission, per the International Working Group Response Criteria for MDS, recorded before and including the first event of progression (treatment failure, relapse after CR or PR, disease transformation, and PD) based on altering the natural history of the disease. Complete remission: <5% bone marrow blasts without evidence of dysplasia; peripheral blood counts: hemoglobin ≥11 grams per deciliter (g/dL), neutrophils ≥1 x 10^9/L, platelets ≥100 x 10^9/L. Partial remission: meeting complete remission criteria, but bone marrow blasts decreased by ≥50% from pre-treatment, but still ≥5%. Bone marrow complete remission: ≤5% bone marrow blasts and decrease by ≥50% from pre-treatment.
Time Frame: up to 61 days
Population: Full Analysis Set. Only participants with MDS who received monotherapy were analyzed. The participant in Group A receiving 3 mg QOD was on treatment for less than a week and therefore was not evaluated for efficacy.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: INCB059872 Monotherapy; 2 mg QOD | Group A: INCB059872 Monotherapy; 2 mg QD | Group A: INCB059872 Monotherapy; 3 mg QOD | Group A: INCB059872 Monotherapy; 3 mg QD | Group A: INCB059872 Monotherapy; 4 mg QD | Group A: INCB059872 Monotherapy; 5 mg QD | Group B: INCB059872 Monotherapy; 1 mg QD | Group B: INCB059872 Monotherapy; 2 mg QOD | Group B: INCB059872 Monotherapy; 2 mg QD | Group B: INCB059872 Monotherapy; 3 mg QOD | Group B: INCB059872 Monotherapy; 3 mg QD | Group B: INCB059872 Monotherapy; 4 mg QOD
Number analyzed (Participants) | 0 | 1 | 0 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
percentage of participants |  | 0.0 |  | 0.0 | 0.0 |  |  |  |  |  |  |

6. Secondary Outcome: Change From Baseline in Spleen Volume Reduction (SVR) at Week 12 in Participants With Myelofibrosis (MF) Who Received INCB059872 Monotherapy
Description: Change from Baseline was to have been calculated as the post-Baseline value minus the Baseline value. SVR was to have been measured by magnetic resonance imaging (MRI), or by computed tomography (CT) scan in participants who were not candidates for MRI or when MRI was not readily available.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Analysis was not conducted because no participants with MF remained in the study at Week 12.
Arm/Group | Group A: INCB059872 Monotherapy; 2 mg QOD | Group A: INCB059872 Monotherapy; 2 mg QD | Group A: INCB059872 Monotherapy; 3 mg QOD | Group A: INCB059872 Monotherapy; 3 mg QD | Group A: INCB059872 Monotherapy; 4 mg QD | Group A: INCB059872 Monotherapy; 5 mg QD | Group B: INCB059872 Monotherapy; 1 mg QD | Group B: INCB059872 Monotherapy; 2 mg QOD | Group B: INCB059872 Monotherapy; 2 mg QD | Group B: INCB059872 Monotherapy; 3 mg QOD | Group B: INCB059872 Monotherapy; 3 mg QD | Group B: INCB059872 Monotherapy; 4 mg QOD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Cmax of INCB059872 in Plasma When Received as Monotherapy
Description: Cmax was defined as the maximum observed plasma concentration of INCB059872.
Time Frame: Cycle 1 Day 15: 0.5, 1, 2, 4, and 6 hours after INCB059872 dose
Population: Pharmacokinetic (PK)-Evaluable Population: all participants who received at least 1 dose of study treatment and provided at least 1 postdose PK sample
Measure: Mean (Standard Deviation); unit: nanomolar (nM)
Arm/Group | Group A: INCB059872 Monotherapy; 2 mg QOD | Group A: INCB059872 Monotherapy; 2 mg QD | Group A: INCB059872 Monotherapy; 3 mg QOD | Group A: INCB059872 Monotherapy; 3 mg QD | Group A: INCB059872 Monotherapy; 4 mg QD | Group A: INCB059872 Monotherapy; 5 mg QD | Group B: INCB059872 Monotherapy; 1 mg QD | Group B: INCB059872 Monotherapy; 2 mg QOD | Group B: INCB059872 Monotherapy; 2 mg QD | Group B: INCB059872 Monotherapy; 3 mg QOD | Group B: INCB059872 Monotherapy; 3 mg QD | Group B: INCB059872 Monotherapy; 4 mg QOD
Number analyzed (Participants) | 2 | 4 | 0 | 3 | 3 | 1 | 3 | 3 | 0 | 6 | 1 | 3
nanomolar (nM) | 33.4 (29.2) | 46.0 (12.5) |  | 73.1 (30.5) | 110 (13.7) | NA (NA) — To protect participant privacy and mitigate the risk of re-identification, mean (SD) cannot be reported for a single participant. | 25.7 (21.8) | 46.0 (9.95) |  | 70.6 (25.6) | NA (NA) — To protect participant privacy and mitigate the risk of re-identification, mean (SD) cannot be reported for a single participant. | 98.2 (28.5)

8. Secondary Outcome: Tmax of INCB059872 in Plasma When Received as Monotherapy
Description: tmax was defined as the time to the maximum observed plasma concentration of INCB059872.
Time Frame: Cycle 1 Day 15: 0.5, 1, 2, 4, and 6 hours after INCB059872 dose
Population: Pharmacokinetic (PK)-Evaluable Population
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: INCB059872 Monotherapy; 2 mg QOD | Group A: INCB059872 Monotherapy; 2 mg QD | Group A: INCB059872 Monotherapy; 3 mg QOD | Group A: INCB059872 Monotherapy; 3 mg QD | Group A: INCB059872 Monotherapy; 4 mg QD | Group A: INCB059872 Monotherapy; 5 mg QD | Group B: INCB059872 Monotherapy; 1 mg QD | Group B: INCB059872 Monotherapy; 2 mg QOD | Group B: INCB059872 Monotherapy; 2 mg QD | Group B: INCB059872 Monotherapy; 3 mg QOD | Group B: INCB059872 Monotherapy; 3 mg QD | Group B: INCB059872 Monotherapy; 4 mg QOD
Number analyzed (Participants) | 2 | 4 | 0 | 3 | 3 | 1 | 3 | 3 | 0 | 6 | 1 | 3
hours | 0.5 [0.5 to 0.5] | 1 [0.5 to 1] |  | 1 [0.5 to 1] | 0.5 [0.5 to 1] | NA [NA to NA] — To protect participant privacy and mitigate the risk of re-identification, median (full range) cannot be reported for a single participant. | 2.0 [0.5 to 2] | 2 [0.5 to 2] |  | 1 [0.5 to 2] | NA [NA to NA] — To protect participant privacy and mitigate the risk of re-identification, median (full range) cannot be reported for a single participant. | 0.5 [0.5 to 1]

9. Secondary Outcome: AUC(0-τ) of INCB059872 in Plasma When Received as Monotherapy
Description: AUC(0-τ) was defined as the area under the plasma concentration-time curve from time = 0 to the end of the dosing period of INCB059872.
Time Frame: Cycle 1 Day 15: 0.5, 1, 2, 4, and 6 hours after INCB059872 dose
Population: Pharmacokinetic (PK)-Evaluable Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nM x hour
Arm/Group | Group A: INCB059872 Monotherapy; 2 mg QOD | Group A: INCB059872 Monotherapy; 2 mg QD | Group A: INCB059872 Monotherapy; 3 mg QOD | Group A: INCB059872 Monotherapy; 3 mg QD | Group A: INCB059872 Monotherapy; 4 mg QD | Group A: INCB059872 Monotherapy; 5 mg QD | Group B: INCB059872 Monotherapy; 1 mg QD | Group B: INCB059872 Monotherapy; 2 mg QOD | Group B: INCB059872 Monotherapy; 2 mg QD | Group B: INCB059872 Monotherapy; 3 mg QOD | Group B: INCB059872 Monotherapy; 3 mg QD | Group B: INCB059872 Monotherapy; 4 mg QOD
Number analyzed (Participants) | 2 | 4 | 0 | 3 | 3 | 1 | 1 | 1 | 0 | 6 | 1 | 3
nM x hour | 196 (8.38) | 216 (75.5) |  | 374 (120) | 486 (107) | NA (NA) — To protect participant privacy and mitigate the risk of re-identification, mean (SD) cannot be reported for a single participant. | NA (NA) — To protect participant privacy and mitigate the risk of re-identification, mean (SD) cannot be reported for a single participant. | NA (NA) — To protect participant privacy and mitigate the risk of re-identification, mean (SD) cannot be reported for a single participant. |  | 361 (115) | NA (NA) — To protect participant privacy and mitigate the risk of re-identification, mean (SD) cannot be reported for a single participant. | 495 (63.2)

10. Secondary Outcome: t1/2 of INCB059872 in Plasma When Received as Monotherapy
Description: t1/2 was defined as the half-life of INCB059872.
Time Frame: Cycle 1 Day 15: 0.5, 1, 2, 4, and 6 hours after INCB059872 dose
Population: Pharmacokinetic (PK)-Evaluable Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group A: INCB059872 Monotherapy; 2 mg QOD | Group A: INCB059872 Monotherapy; 2 mg QD | Group A: INCB059872 Monotherapy; 3 mg QOD | Group A: INCB059872 Monotherapy; 3 mg QD | Group A: INCB059872 Monotherapy; 4 mg QD | Group A: INCB059872 Monotherapy; 5 mg QD | Group B: INCB059872 Monotherapy; 1 mg QD | Group B: INCB059872 Monotherapy; 2 mg QOD | Group B: INCB059872 Monotherapy; 2 mg QD | Group B: INCB059872 Monotherapy; 3 mg QOD | Group B: INCB059872 Monotherapy; 3 mg QD | Group B: INCB059872 Monotherapy; 4 mg QOD
Number analyzed (Participants) | 2 | 4 | 0 | 3 | 3 | 1 | 1 | 1 | 0 | 6 | 1 | 3
hours | 3.15 (0.189) | 3.30 (0.765) |  | 3.13 (0.495) | 3.67 (1.38) | NA (NA) — To protect participant privacy and mitigate the risk of re-identification, mean (SD) cannot be reported for a single participant. | NA (NA) — To protect participant privacy and mitigate the risk of re-identification, mean (SD) cannot be reported for a single participant. | NA (NA) — To protect participant privacy and mitigate the risk of re-identification, mean (SD) cannot be reported for a single participant. |  | 3.57 (0.52) | NA (NA) — To protect participant privacy and mitigate the risk of re-identification, mean (SD) cannot be reported for a single participant. | 4.28 (0.25)

11. Secondary Outcome: CL/F of INCB059872 in Plasma When Received as Monotherapy
Description: CL/F was defined as the apparent oral clearance of INCB059872.
Time Frame: Cycle 1 Day 15: 0.5, 1, 2, 4, and 6 hours after INCB059872 dose
Population: Pharmacokinetic (PK)-Evaluable Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Group A: INCB059872 Monotherapy; 2 mg QOD | Group A: INCB059872 Monotherapy; 2 mg QD | Group A: INCB059872 Monotherapy; 3 mg QOD | Group A: INCB059872 Monotherapy; 3 mg QD | Group A: INCB059872 Monotherapy; 4 mg QD | Group A: INCB059872 Monotherapy; 5 mg QD | Group B: INCB059872 Monotherapy; 1 mg QD | Group B: INCB059872 Monotherapy; 2 mg QOD | Group B: INCB059872 Monotherapy; 2 mg QD | Group B: INCB059872 Monotherapy; 3 mg QOD | Group B: INCB059872 Monotherapy; 3 mg QD | Group B: INCB059872 Monotherapy; 4 mg QOD
Number analyzed (Participants) | 2 | 4 | 0 | 3 | 3 | 1 | 1 | 1 | 0 | 6 | 1 | 3
Liters per hour | 32.9 (7.94) | 26.3 (9.31) |  | 22.1 (6.56) | 22.1 (5.57) | NA (NA) — To protect participant privacy and mitigate the risk of re-identification, mean (SD) cannot be reported for a single participant. | NA (NA) — To protect participant privacy and mitigate the risk of re-identification, mean (SD) cannot be reported for a single participant. | NA (NA) — To protect participant privacy and mitigate the risk of re-identification, mean (SD) cannot be reported for a single participant. |  | 23.1 (6.32) | NA (NA) — To protect participant privacy and mitigate the risk of re-identification, mean (SD) cannot be reported for a single participant. | 21.1 (2.74)

12. Secondary Outcome: ORR in Participants With SCLC Who Received Combination Therapy
Description: ORR was defined as the percentage of participants who achieved a best overall response of CR or a PR, per investigator assessment according to RESIST v1.1, recorded before and including the first event of PD. CR: disappearance of all target and non-target lesions and no appearance of any new lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to <10 mm. PR: complete disappearance or at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum diameters, no new lesions, and no progression of non-target lesions.
Time Frame: up to 1353 days
Population: Full Analysis Set. Only participants with SCLC who received combination therapy and had available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5
percentage of participants |  |  |  |  |  | 20.0

13. Secondary Outcome: ORR for Altering the Natural History of the Disease in Participants With AML Who Received Combination Therapy
Description: ORR was defined as the percentage of participants who achieved a best overall response of complete remission or CRi, per the International Working Group Response Criteria for AML, recorded before and including the first event of progression (treatment failure, relapse, and PD) based on altering the natural history of the disease. Complete remission: ANC ≥1.0 x 10^9/L, platelet count ≥100 x 10^9/L, bone marrow with less than 5% blast cells, Auer rods not detectable; no platelet, or whole blood transfusions for 7 days prior to the date of the hematology assessment. CRi: complete remission, but the ANC count may be < 1.0 x 10^9/L and/or the platelet count may be <100 x 10^9/L.
Time Frame: up to 208 days
Population: Full Analysis Set. Only participants with AML who received combination therapy were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab
Number analyzed (Participants) | 5 | 7 | 1 | 6 | 1 | 0
percentage of participants | 20.0 | 0.0 | 0.0 | 16.7 | 0.0 |

14. Secondary Outcome: ORR for Altering the Natural History of the Disease in Participants With MDS Who Received Combination Therapy
Description: ORR was defined as the percentage of participants who achieved a best overall response of complete remission, partial remission, or bone marrow complete remission, per the International Working Group Response Criteria for MDS, recorded before and including the first event of progression (treatment failure, relapse after CR or PR, disease transformation, and PD) based on altering the natural history of the disease. Complete remission: <5% bone marrow blasts without evidence of dysplasia; peripheral blood counts: hemoglobin ≥11 g/dL, neutrophils ≥1 x 10^9/L, platelets ≥100 x 10^9/L. Partial remission: meeting complete remission criteria, but bone marrow blasts decreased by ≥50% from pre-treatment, but still ≥5%. Bone marrow complete remission: ≤5% bone marrow blasts and decrease by ≥50% from pre-treatment.
Time Frame: up to 85 days
Population: Full Analysis Set. Only participants with MDS who received combination therapy were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0
percentage of participants |  |  |  | 0.0 |  |

15. Secondary Outcome: Cmax of INCB059872 in Plasma When Received as Combination Therapy
Description: Cmax was defined as the maximum observed plasma concentration of INCB059872.
Time Frame: Cycle 1 Day 15: 0.5, 1, 2, 4, and 6 hours after INCB059872 dose
Population: PK-Evaluable Population
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab
Number analyzed (Participants) | 4 | 2 | 0 | 3 | 0 | 5
nM | 44.3 (16.4) | 96.4 (10.7) |  | 38.2 (33.5) |  | 78.0 (26.3)

16. Secondary Outcome: Tmax of INCB059872 in Plasma When Received as Combination Therapy
Description: tmax was defined as the time to the maximum observed plasma concentration of INCB059872.
Time Frame: Cycle 1 Day 15: 0.5, 1, 2, 4, and 6 hours after INCB059872 dose
Population: PK-Evaluable Population
Measure: Median (Full Range); unit: hours
Arm/Group | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab
Number analyzed (Participants) | 4 | 2 | 0 | 3 | 0 | 5
hours | 1.0 [0.5 to 1] | 0.5 [0.5 to 0.5] |  | 0.5 [0 to 1] |  | 1.0 [0.5 to 1]

17. Secondary Outcome: AUC(0-τ) of INCB059872 in Plasma When Received as Combination Therapy
Description: as for outcome 9
Time Frame: Cycle 1 Day 15: 0.5, 1, 2, 4, and 6 hours after INCB059872 dose
Population: PK-Evaluable Population
Measure: Mean (Standard Deviation); unit: nM x hour
Arm/Group | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab
Number analyzed (Participants) | 4 | 2 | 0 | 3 | 0 | 5
nM x hour | 225 (85.9) | 377 (25.7) |  | 273 (24.4) |  | 357 (97.5)

18. Secondary Outcome: t1/2 of INCB059872 in Plasma When Received as Combination Therapy
Description: t1/2 was defined as the half-life of INCB059872.
Time Frame: Cycle 1 Day 15: 0.5, 1, 2, 4, and 6 hours after INCB059872 dose
Population: PK-Evaluable Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab
Number analyzed (Participants) | 4 | 2 | 0 | 3 | 0 | 5
hours | 3.95 (0.499) | 3.41 (0.281) |  | 3.08 (0.040) |  | 3.79 (0.852)

19. Secondary Outcome: CL/F of INCB059872 in Plasma When Received as Combination Therapy
Description: CL/F was defined as the apparent oral clearance of INCB059872.
Time Frame: Cycle 1 Day 15: 0.5, 1, 2, 4, and 6 hours after INCB059872 dose
Population: PK-Evaluable Population
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab
Number analyzed (Participants) | 4 | 2 | 0 | 3 | 0 | 5
Liters per hour | 25.1 (7.21) | 20.7 (1.41) |  | 19.0 (1.70) |  | 23.5 (8.14)

ADVERSE EVENTS:
Time Frame: up to 1387 days
Description: Treatment-emergent adverse events, defined as adverse events either reported for the first time or the worsening of pre-existing events after the first dose of study drug and within 30 days of the last administration of study drug, have been reported for the Safety Population.
Arm/Group | Group A: INCB059872 Monotherapy; 2 mg QOD | Group A: INCB059872 Monotherapy; 2 mg QD | Group A: INCB059872 Monotherapy; 3 mg QOD | Group A: INCB059872 Monotherapy; 3 mg QD | Group A: INCB059872 Monotherapy; 4 mg QD | Group A: INCB059872 Monotherapy; 5 mg QD | Group B: INCB059872 Monotherapy; 1 mg QD | Group B: INCB059872 Monotherapy; 2 mg QOD | Group B: INCB059872 Monotherapy; 2 mg QD | Group B: INCB059872 Monotherapy; 3 mg QOD | Group B: INCB059872 Monotherapy; 3 mg QD | Group B: INCB059872 Monotherapy; 4 mg QOD | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab
All-Cause Mortality (participants affected / at risk) | 2/3 | 5/6 | 0/1 | 4/5 | 15/18 | 2/2 | 3/3 | 3/3 | 0/1 | 27/36 | 2/3 | 5/7 | 5/5 | 6/7 | 1/1 | 3/7 | 1/1 | 3/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 5/6 | 0/1 | 3/5 | 10/18 | 2/2 | 2/3 | 1/3 | 1/1 | 24/36 | 2/3 | 3/7 | 4/5 | 4/7 | 0/1 | 6/7 | 1/1 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 1/1 | 5/5 | 17/18 | 2/2 | 3/3 | 3/3 | 1/1 | 35/36 | 3/3 | 7/7 | 4/5 | 7/7 | 1/1 | 7/7 | 1/1 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: INCB059872 Monotherapy; 2 mg QOD (N=3) | Group A: INCB059872 Monotherapy; 2 mg QD (N=6) | Group A: INCB059872 Monotherapy; 3 mg QOD (N=1) | Group A: INCB059872 Monotherapy; 3 mg QD (N=5) | Group A: INCB059872 Monotherapy; 4 mg QD (N=18) | Group A: INCB059872 Monotherapy; 5 mg QD (N=2) | Group B: INCB059872 Monotherapy; 1 mg QD (N=3) | Group B: INCB059872 Monotherapy; 2 mg QOD (N=3) | Group B: INCB059872 Monotherapy; 2 mg QD (N=1) | Group B: INCB059872 Monotherapy; 3 mg QOD (N=36) | Group B: INCB059872 Monotherapy; 3 mg QD (N=3) | Group B: INCB059872 Monotherapy; 4 mg QOD (N=7) | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA (N=5) | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA (N=7) | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA (N=1) | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine (N=7) | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine (N=1) | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal haemorrhage (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 6 (8) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: INCB059872 Monotherapy; 2 mg QOD (N=3) | Group A: INCB059872 Monotherapy; 2 mg QD (N=6) | Group A: INCB059872 Monotherapy; 3 mg QOD (N=1) | Group A: INCB059872 Monotherapy; 3 mg QD (N=5) | Group A: INCB059872 Monotherapy; 4 mg QD (N=18) | Group A: INCB059872 Monotherapy; 5 mg QD (N=2) | Group B: INCB059872 Monotherapy; 1 mg QD (N=3) | Group B: INCB059872 Monotherapy; 2 mg QOD (N=3) | Group B: INCB059872 Monotherapy; 2 mg QD (N=1) | Group B: INCB059872 Monotherapy; 3 mg QOD (N=36) | Group B: INCB059872 Monotherapy; 3 mg QD (N=3) | Group B: INCB059872 Monotherapy; 4 mg QOD (N=7) | Group C: Combination Therapy; INCB059872 2 mg QD + ATRA (N=5) | Group C: Combination Therapy; INCB059872 3 mg QD + ATRA (N=7) | Group C: Combination Therapy; INCB059872 4 mg QD + ATRA (N=1) | Group D: Combination Therapy; INCB059872 2 mg QD + Azacitidine (N=7) | Group D: Combination Therapy; INCB059872 3 mg QD + Azacitidine (N=1) | Group E: Combination Therapy; INCB059872 3 mg QOD + Nivolumab (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 8 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial enlargement (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 7 (8) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 6 (6) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 17 (19) | 2 (3) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 5 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival hypertrophy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 10 (10) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral blood blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 7 (8) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 2 (5) | 4 (5) | 0 (0) | 1 (2) | 0 (0) | 5 (12) | 0 (0) | 3 (6)
Tongue haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated by the sponsor due to a strategic business decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT02712905/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT02712905/SAP_001.pdf